CLINICAL TRIAL: NCT07143578
Title: Comparison Of Surgical Management Of Early Pregnancy Loss By Suction Curettage Versus Hysteroscopy In Patients Undergoing In-Vitro Fertilization (IVF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Noam Smorgick, Director of MIGS, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0162-25-ASF
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Early Abortion; Pregnancy Loss, Early
Keywords: hysteroscopy; pregnancy loss; early missed abortion; spontaneous abortion; suction curettage; intrauterine adhesions
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Missed; Gynatresia | interventions — Vacuum Curettage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operative hysteroscopy (Experimental): Operative hysteroscopy using tissue removal device
  Interventions: Device: Operative hysteroscopy using tissue removal device
- Suction curretage (Active Comparator): Standard suction curettage
  Interventions: Device: suction curettage

INTERVENTIONS:
Device: Operative hysteroscopy using tissue removal device — Operative hysteroscopy using tissue removal device
  Arms: Operative hysteroscopy
Device: suction curettage — suction curettage using plastic scution curette
  Arms: Suction curretage

SUMMARY:
Early pregnancy loss occurs in ~15% of pregnancies. The treatment options include surgical uterine evacuation by suction curettage, medical management with misoprostol, or conservative management without interventions. The advantages of surgical management include quick resolution of the pregnancy and avoidance of heavy vaginal bleeding, while the disadvantages include retained products of conception and intrauterine adhesion formation which could affect future fertility. With the aim of reducing the complications of suction curettage, uterine evacuation using operative hysteroscopy has been suggested.

In a previous study, the investigators compared suction curettage with operative hysteroscopy for the surgical management of early pregnancy loss up to 10 weeks of gestation. The results showed significantly reduced adhesions rate (4.2% in the hysteroscopy group vs. 45.2% in the suction group, p < 0.01), although the operative time was significantly longer for the hysteroscopy.

In this follow-up study, the investigators will compare the outcomes of hysteroscopy and suction curettage in a select group of patients with early pregnancy loss following conception by in-vitro fertilization. These patients are at risk for adhesions and therefore candidates for the hysteroscopic intervention. The study will include 50 patients randomized to 2 intervention arms - hysteroscopy using a tissue removal device versus the standard suction curettage. Post-operative adhesions will be assessed by office hysteroscopy after 6-8 weeks.

DETAILED DESCRIPTION:
The treatment options for early pregnancy loss include surgical uterine evacuation by suction curettage, medical management with misoprostol, and expectant (conservative) management. The advantages of surgical evacuation include quick resolution of the pregnancy and prevention of heavy bleeding that could necessitate urgent curettage. Although suction curettage is a common and relatively safe procedure, it carries short term risks such as infection, retained products of conception requiring repeat surgery, hemorrhage, and uterine perforation. Long term complications include intrauterine adhesions (also known as Asherman's syndrome), which may impair fertility. In recent years, the option of uterine evacuation by operative hysteroscopy has been investigated. Hysteroscopy enables a visual inspection of the uterine cavity (as opposed to the blind suction curettage), and involves a targeted and limited contact with the endometrium, possibly reducing adhesion formation compared to the "global" suction curettage.

Previous studies indeed found that hysteroscopy was feasible and safe for the surgical management of early pregnancy loss. The investigators recently completed a prospective RCT comparing suction curettage and operative hysteroscopy in 100 women diagnosed with early pregnancy loss up to 10 weeks of gestation. The results showed a significantly lower rate of intrauterine adhesions in the hysteroscopy group (4.2% vs. 45.2%, p < 0.01). However, operative time was significantly longer for the hysteroscopy. There were no significant differences between groups in the rates of retained products of conception or surgical complications.

Although the study did not address the cost of the different surgical techniques, hysteroscopy is obviously more expensive and requires specialized equipment and skilled surgeons. Thus, operative hysteroscopy is likely more applicable for selected patients at risk for intrauterine adhesions and impaired fertility.

Patients undergoing in-vitro fertilization (UVF) represent a unique population with higher baseline risk for intrauterine adhesions due to prior uterine procedures and repeated curettage. Hooker et al. demonstrated that adhesions could cause impair embryo implantation, thereby reducing the rate of successful IVF cycles. Deng et al. showed that delaying embryo transfer after adhesiolysis improves live birth rates.

In view of the impact of adhesions on fertility and the potential to delay pregnancy, selecting the optimal surgical method is especially important for IVF patients diagnosed with early pregnancy loss, and these patients may benefit specifically from the hysteroscopic procedure.

This study is a randomized controlled, non-blinded study interventional study comparing operative hysteroscopy and suction curettage for the surgical management of early pregnancy loss in patients undergoing in-vitro fertilization. The study will include 50 patients (25 in each arm) diagnosed with early pregnancy loss ≤10 weeks. The study will compare procedural feasibility, safety, postoperative intrauterine adhesions and retained products of conception, as well as time to the next pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of early pregnancy loss up to 10 weeks' gestation, based on last menstrual period or ultrasound.
2. Pregnancy conceived through assisted reproductive techniques (in vitro fertilization, IVF).
3. Ability to provide informed consent, and proficiency in reading and writing Hebrew.

Exclusion Criteria:

1. Heavy vaginal bleeding or diagnosis of incomplete abortion.
2. Signs of infection and/or suspicion of septic abortion
3. Known uterine anomalies- including septate, bicornuate, unicornuate, or didelphys uterus.
4. Prior medical or surgical treatment during the current pregnancy
5. History of intrauterine adhesions
6. History of ≥ 3 prior miscarriages.
7. History of ≥ 3 prior cesarean sections.
8. History of myomectomy via abdominal or hysteroscopic approach.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Individuals who can carry a pregnancy
Enrollment: 50 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Intrauterine adhesions | 8 weeks
  Post-operative intrauterine adhesions will be evaluated by office diagnostic hysteroscopy after 6-8 weeks. The physician performing the office hysteroscopy will be blinded to the patient's intervention arm. The intrauterine adhesions will be classified according to the American Fertility Society score (from 0 to 12, higher scores means worse adhesions).
Time to pregnancy | 12 months
  The patient's reproductive outcomes will be assessed by telephone interview after 6 and 12 months from the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Smorgick, MD, Principal Investigator — Assaf-Harofeh Medical Center; Maya Naor Dovev, MD, Study Director — Assaf-Harofeh Medical Center
Locations (2):
- Israel (2):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Sheba Medical Center, Tel Hashomer, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huchon C, Drioueche H, Koskas M, Agostini A, Bauville E, Bourdel N, Fernandez H, Fritel X, Graesslin O, Legendre G, Lucot JP, Panel P, Raiffort C, Giraudet G, Bussieres L, Fauconnier A. Operative Hysteroscopy vs Vacuum Aspiration for Incomplete Spontaneous Abortion: A Randomized Clinical Trial. JAMA. 2023 Apr 11;329(14):1197-1205. doi: 10.1001/jama.2023.3415. PMID 37039805
- [Background] Bar-On S, Berkovitz Shperling R, Cohen A, Akdam A, Michaan N, Levin I, Rattan G, Tzur Y. Primary Resectoscopic Treatment of First-Trimester Miscarriage. J Obstet Gynaecol Can. 2024 Apr;46(4):102327. doi: 10.1016/j.jogc.2023.102327. Epub 2023 Dec 1. PMID 38042480
- [Background] Quenby S, Gallos ID, Dhillon-Smith RK, Podesek M, Stephenson MD, Fisher J, Brosens JJ, Brewin J, Ramhorst R, Lucas ES, McCoy RC, Anderson R, Daher S, Regan L, Al-Memar M, Bourne T, MacIntyre DA, Rai R, Christiansen OB, Sugiura-Ogasawara M, Odendaal J, Devall AJ, Bennett PR, Petrou S, Coomarasamy A. Miscarriage matters: the epidemiological, physical, psychological, and economic costs of early pregnancy loss. Lancet. 2021 May 1;397(10285):1658-1667. doi: 10.1016/S0140-6736(21)00682-6. Epub 2021 Apr 27. PMID 33915094